CLINICAL TRIAL: NCT06298227
Title: The Comparison of Erector Spinae Plane Block and Quadratus Lumborum Block on Postoperative Analgesia in Patients Undergoing Laparoscopic Nephrectomy: A Randomized, Prospective, Controlled Study
Brief Title: Erector Spinae Plane Block vs Quadratus Lumborum Block for Laparoscopic Nephrectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, Ayse Ince, Principal Investigator, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Medipol Hospital 1
Record Dates: First submitted 2024-02-06; First posted 2024-03-07 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Kidney Diseases; Kidney Failure
Keywords: Laparoscopic nephrectomy; Postoperative pain management; Erector spinae plane block; Quadratus lumborum block
MeSH Terms: conditions — Kidney Diseases; Renal Insufficiency | interventions — Analgesia, Patient-Controlled

STUDY DESIGN:
Intervention Model Description: Sixty patients aged 18-65 years old with American Society of Anesthesiologists (ASA) classification I-II and scheduled for laparoscopic nephrectomy surgery will be included in the study. Patients will be randomly divided into two groups (Group ESPB = ESPB group, Group QLB = QLB group) including 30 patients each, before entering the operating room.
Who Masked: Participant, Outcomes Assessor
Masking Description: Outcomes assessor and participants will be blinded to the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group ESPB = Erector spinae plane block group (Active Comparator): ESPB will be performed
  Interventions: Other: Postoperative analgesia management with Paracerol® and IV PCA with Talinat®; Other: Erector spinae plane block
- Group QLB = Quadratus lumborum block group (Active Comparator): QLB will be performed
  Interventions: Other: Postoperative analgesia management with Paracerol® and IV PCA with Talinat®; Other: Quadratus lumborum plane block

INTERVENTIONS:
Other: Postoperative analgesia management with Paracerol® and IV PCA with Talinat® — In the postoperative period, 1 g of acetaminophen (Paracerol®) will be administered intravenously to patients every 8 hours. Patients in all groups will have IV patient-controlled analgesia (PCA- CADD-Solis®) containing 10 mcg/ml fentanyl ( Talinat®). 10 mcg bolus without infusion dose, 20-minute lock time will be the protocol. Postoperative patient evaluation will be performed by another anesthesiologist. If the NRS score is ≥ 4, 0.5 mg/kg IV meperidine (Aldolan®) will be administered as a rescue analgesic.
Other: Erector spinae plane block — The block will be applied while the patient is in the lateral decubitus position. The convex probe of US ( GE Healthcare®) will be placed longitudinally 4 cm lateral to the T11 transverse process. The erector spinae muscle and the hyperechoic transverse process will be visualized. Using the in-plane technique, the 100 mm block needle (Stimuplex 360®) will be advanced in the cranio-caudal direction and 5 ml of saline will be injected under the erector spinae muscle to confirm the block location. Once the block location is confirmed, 40 ml of 0.25% bupivacaine (Marcaine®) will be administered.
  Arms: Group ESPB = Erector spinae plane block group
Other: Quadratus lumborum plane block — QLB will be performed with the patient in the lateral decubitus position. The convex probe of US ( GE Healthcare®) will be placed at the level of the 12th rib, just above the iliac crest, in the parasagittal oblique plane, at the L1-L2 level. After the quadratus lumborum, erector spinae, and psoas major muscles are visualized, a 100 mm block needle (Stimuplex 360®) will be advanced in-plane anteriorly to QL, and the needle tip will be brought between the QL and PM muscles (Anterior QLB). The location will be confirmed by hydraulic dissection with 5 ml saline injection. After the block location is confirmed, 40 ml of 0.25% bupivacaine (Marcaine®) will be administered.
  Arms: Group QLB = Quadratus lumborum block group

SUMMARY:
Ultrasound (US) guided Quadratus Lumborum Block (QLB) is performed at the level of the 12th rib, in the parasagittal oblique plane, at the L1-L2 level. As there are modifications of the block generally local anesthetic is given between quadratus lumborum (QL) and psoas major (PM) muscles (Anterior QLB). The QLB provides a sensory block between T7 - L1. Therefore, QLBs are used to provide postoperative analgesia for abdominal, obstetric, gynecologic, and urologic surgeries.

US-guided erector spinae plane block (ESPB) is performed at the level of the T11 transverse process. After visualization of the erector spinae (ES) muscle and the transverse process, local anesthetic is injected under the ES muscle. ESPB provides a sensory block of the anterior, posterior, and lateral thoracic and abdominal walls accordingly it's used for postoperative analgesia after thoracal wall repairs, thoracotomies, percutaneous nephrolithotomies, nephrectomies, and ventral hernia repairs.

This study aims to compare the effectiveness of US-guided ESPB and QLB on postoperative pain control after laparoscopic nephrectomy.

DETAILED DESCRIPTION:
Nephrectomy for renal transplantation is a commonly performed procedure. The laparoscopic live donor nephrectomy (LLDN) is associated with many benefits and has become the gold standard for kidney retrieval surgery. As compared to open donor nephrectomy (ODN), LLDN has been shown to have less post-operative pain, shorter hospital stays, and faster recovery. Even though LLDN is less traumatic, some patients undergoing laparoscopic live donor nephrectomy still suffer significant postoperative pain require parenteral opioids, and have a risk for chronic pain.

The postoperative pain mechanism of LLDN is multifactorial - port pain, pain caused by incisions to retrieve the kidney, pelvic organ nociception, diaphragmatic irritation, and discomfort of a urinary catheter. Opioids, epidural anesthesia, Transversus Abdominal Plane (TAP) Block, and local infiltration of local anesthetics are used to prevent postoperative pain after LLDN.

In this study, the investigators aim to compare the effectiveness of US-guided ESPB and QLB on postoperative pain control after laparoscopic nephrectomy.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) classification I-II
* Scheduled for living donor laparoscopic nephrectomy under general anesthesia

Exclusion Criteria:

* history of bleeding diathesis,
* receiving anticoagulant treatment,
* known local anesthetics and opioid allergy,
* infection of the skin at the site of the needle puncture,
* pregnancy or lactation,
* patients who refuse the procedure or participation in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-03-11 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Amount of total opioid consumption (Fentanyl PCA) at the first 24 hours period postoperatively | Changes from baseline opioid consumption at postoperative 1, 2, 4, 8, 16 and 24 hours.
  The primary aim is to compare postoperative opioid consumption from the PCA device.

SECONDARY OUTCOMES:
Pain scores (Numerical rating scale-NRS) | Changes from baseline pain scores at postoperative 1, 2, 4, 8, 16 and 24 hours
  The secondary aim is to compare NRS at the postoperative 24 h. Postoperative pain assessment will be performed using the NRS (0 = no pain, 10 = the most severe pain felt). The NRS scores will be recorded
Need for rescue analgesia (meperidine) | Postoperative 24 hours period
  The secondary aim is to compare rescue analgesia used in the postoperative 24 h.
Adverse events | Postoperative 24 hours period
  The secondary aim is to compare the adverse events (nausea, vomiting, itching) related to opioid use.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University Mega Hospital Complex, Istanbul, Bağcılar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The investigators will not share individual patient data(IPD)

REFERENCES:
- [Background] Elsharkawy H, Ahuja S, Sessler DI, Maheshwari K, Mao G, Sakr Esa WA, Soliman LM, Ayad S, Khoshknabi D, Khan MZ, Raza S, DeGrande S, Turan A. Subcostal Anterior Quadratus Lumborum Block Versus Epidural Block for Analgesia in Open Nephrectomy: A Randomized Clinical Trial. Anesth Analg. 2021 Apr 1;132(4):1138-1145. doi: 10.1213/ANE.0000000000005382. PMID 33617181
- [Background] Alvi AS, Nasir JA, Nizam MA, Hamdani MM, Bhangar NA, Sibtain SA, Lalani AS, Warle MC. Quadratus lumborum block and transversus abdominis plane block in laparoscopic nephrectomy: a meta-analysis. Pain Manag. 2023 Sep;13(9):555-567. doi: 10.2217/pmt-2023-0033. Epub 2023 Sep 18. PMID 37718911
- [Background] Wang J, Chu T, Sun R, Xu A. Analgesic Efficacy of Quadratus Lumborum Block in Patients Undergoing Nephrectomy: A Systematic Review and Meta-Analysis. Pain Med. 2023 May 2;24(5):476-487. doi: 10.1093/pm/pnac166. PMID 36321993
- [Background] Sahin A, Baran O. Effect of ultrasound-guided erector spinae plane block on post-surgical pain in patients undergoing nephrectomy: a single-center, randomized, double-blind, controlled trial. J Int Med Res. 2022 Mar;50(3):3000605221086737. doi: 10.1177/03000605221086737. PMID 35301896
- [Background] Fan Q, Liu H, Li Y, Dai H, Wang Y. Comparison of ultrasound-guided erector spinae plane block and thoracic paravertebral block for postoperative analgesia after laparoscopic nephrectomy: a randomized controlled non-inferiority clinical trial. Minerva Anestesiol. 2023 Jun;89(6):520-528. doi: 10.23736/S0375-9393.22.16794-5. Epub 2023 Jan 24. PMID 36692339